CLINICAL TRIAL: NCT01696578
Title: Effectiveness of Combined Intervention Approaches in the Treatment of Affective Disorders and Chronic Pain in Victims of Torture and Massive Violence in Kosovo: A Randomized Controlled Trial
Brief Title: Effectiveness of Combined Intervention Approaches in the Treatment of Affective Disorders and Chronic Pain in War Victims
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehabilitation and Research Centre for Torture Victims (Other)
Collaborators: Kosova Rehabilitation Centre for Torture Victims (Other)
Responsible Party: Principal Investigator, Shr-Jie Wang, Principal investigator, Rehabilitation and Research Centre for Torture Victims
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCTF5S2P4D1
Record Dates: First submitted 2012-09-25; First posted 2012-10-01 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: PTSD; Depression; Anxiety; Chronic Pain; Anger
Keywords: PTSD; Depression; Anxiety; Chronic pain; Anger; Heart rate variability; Disability
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders; Chronic Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BF-CBT and group physiotherapy (Experimental): Multivitamin+10 sessions of biofeedback supported cognitive behavioral therapy (BF-CBT) and 10 sessions of group physiotherapy
  Interventions: Behavioral: BF-CBT and group physiotherapy
- Waiting list (Active Comparator): The waiting list group receives only multivitamin pills while being waiting and will receive the same intervention 3 months later
  Interventions: Behavioral: BF-CBT and group physiotherapy

INTERVENTIONS:
Behavioral: BF-CBT and group physiotherapy — Multivitamin+10 individual therapy sessions (BF-CBT) and 10 group therapy sessions (physical exercises) on a weekly basis

SUMMARY:
This study will measure the effects of biofeedback supported cognitive behavioral therapy (BF-CBT) and group physiotherapy intervention in victims of torture and massive violence in Kosovo. The investigators aim to restore physical and psychosocial functioning of the victims of torture and massive violence with available rehabilitation practice and integrate them into the community. It is also our objective to build local knowledge and expertise to apply measurement principles and CBT methods in the Balkan region.

DETAILED DESCRIPTION:
The primary objective of this project is to contribute to the promotion of evidence-based health intervention which is dealing with the long-term consequences of trauma in the post-conflict Kosovo.

This is the second phase of a series of multi-site case studies. Based on the knowledge generated in the first phase of project in 2007-2009, the investigators conclude that there is a need to continue with health interventions in northern Kosovo among those who are still suffering from the long-term effects of trauma. Many problems need to be addressed, ranging from unemployment and sleep disturbances to a high suicide rate. As our study shows, the situation is frequently complicated by co-morbidity between mental and physical problems, in particular, anger, hatred, severe depression and chronic pain.

At this phase, the investigators aim to provide the available rehabilitation service to the victims of torture and massive violence in northern Kosovo. The investigators undertake an integrated intervention approach; that is a biofeedback supported cognitive-behavioral therapy (BF-CBT), which involves anger management, anxiety and phobia treatment (based on prolong exposure therapy)and a group physiotherapy intervention, which promotes physical fitness and social participation. The ultimate goal of this project is to determine both feasibility and the effectiveness of combined interventions in the countries with limited resources.

ELIGIBILITY:
Inclusion Criteria:

* Victims of massive violence from northern Kosovo who reported one or more of the following experiences: 1) torture and other cruel, inhuman or degrading treatment or punishment (TCIDTP); 2) sexual harassment, molestation, rape or insertion of a blunt object into a genital organ and/or the rectum; 3) arrest and detention without warrant or order; or 4) extrajudicial execution of family members, perpetrated by members of law enforcement agency.
* Clinical diagnosis of PTSD and one of following symptoms: depression, anxiety or chronic pain

Exclusion Criteria:

* With mental retardation or significant speech or cognitive impairment that would impede assessments
* With past or present schizophrenia
* With major alcoholic or substance abuse problems
* Having recently undergone chemotherapy or chemo-radiotherapy for cancer or will have these therapy within following 6 months,
* Having had any CBT in the past three years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change of depression symptom from baseline at 3 and 6 months | 0-3-6 months
Change of anxiety symptom from baseline at 3 and 6 months | 0-3-6 months
Change of chronic pain symptom from baseline at 3 and 6 months | 0-3-6 months
Change of anger from baseline at 3 and 6 months | 0-3-6 months
Change of PTSD symptom from baseline at 3 and 6 months | 0-3-6 months

SECONDARY OUTCOMES:
Change of disability scale from baseline at 3 and 6 months | 0-3-6 months
Change of hand-grip strength from baseline at 3 and 6 months | 0-3-6 months
Change of standing balance from baseline at 3 and 6 months | 0-3-6 months
Change of BMI from baseline at 3 and 6 months | 0-3-6 months
Change of heart rate variability from baseline at 3 and 6 months | 0-3-6 months

OTHER OUTCOMES:
Change of reporting sleep disorder from baseline at 3 and 6 months | 0-3-6 months
Change of reporting suicide ideation from baseline at 3 and 6 months | 0-3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shr-Jie Wang, Ph.D., Principal Investigator — Rehabilitation and Research Centre for Torture Victims
Locations (1):
- Kosova Rehabilitation Centre for Torture Victims, Pristina, Kosovo

REFERENCES:
- [Background] Wang SJ, Salihu M, Rushiti F, Bala L, Modvig J. Survivors of the war in the Northern Kosovo: violence exposure, risk factors and public health effects of an ethnic conflict. Confl Health. 2010 May 28;4:11. doi: 10.1186/1752-1505-4-11. PMID 20509915
- [Background] Wang SJ, Pacolli S, Rushiti F, Rexhaj B, Modvig J. Survivors of war in the Northern Kosovo (II): baseline clinical and functional assessment and lasting effects on the health of a vulnerable population. Confl Health. 2010 Sep 21;4:16. doi: 10.1186/1752-1505-4-16. PMID 20858274
- [Background] Wang SJ, Rushiti F, Sejdiu X, Pacolli S, Gashi B, Salihu F, Modvig J. Survivors of war in northern Kosovo (III): The role of anger and hatred in pain and PTSD and their interactive effects on career outcome, quality of sleep and suicide ideation. Confl Health. 2012 Jul 30;6(1):4. doi: 10.1186/1752-1505-6-4. PMID 22846511
- [Derived] Wang SJ, Bytyci A, Izeti S, Kallaba M, Rushiti F, Montgomery E, Modvig J. A novel bio-psycho-social approach for rehabilitation of traumatized victims of torture and war in the post-conflict context: a pilot randomized controlled trial in Kosovo. Confl Health. 2017 Feb 8;10:34. doi: 10.1186/s13031-016-0100-y. eCollection 2016. PMID 28191034